CLINICAL TRIAL: NCT03046914
Title: A Prospective Study to Prove the Usefulness of HLA-B*5801 Screening Test for the Prevention of Allopurinol-induced Severe Cutaneous Adverse Reaction in Patient With Chronic Kidney Disease
Brief Title: HLA-B*5801 Screening to Prevent Allopurinol-induced Severe Cutaneous Adverse Reaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Heung-Woo Park, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SNUIMA002
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Stevens-Johnson Syndrome; Kidney Failure, Chronic
MeSH Terms: conditions — Stevens-Johnson Syndrome; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective cases and historical controls
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLA-B*5801 screen test (Experimental): An arm in which a participant takes HLA-B*5801 test before administration of allopurinol
  Interventions: Genetic: HLA-B*5801 test

INTERVENTIONS:
Genetic: HLA-B*5801 test — Check whether a participant has HLA-B*5801 allele or not, before administration of allopurinol

SUMMARY:
Allopurinol-induced severe cutaneous adverse reaction (SCAR) is a rare but fatal condition. Previous reports have reported that HLA-B*5801 is an important genetic risk factor significantly associated with the development of allopurinol-induced SCAR. However, there has been no prospective study to prove the clinical efficacy of a HLA-B*5801 screening before administration of allopurinol in predicting allopurinol-induced SCAR. The purpose of this prospective study is to test our hypothesis that a pre-screening of HLA-B*5801 will significantly reduce the risk of allopurinol-induced SCAR development compared to the historical control.

ELIGIBILITY:
Inclusion Criteria:

* a subject who needs an allopurinol treatment based on the physician's assessement
* a subject with chronic kidney disease (CKD)

  * CKD is diagnosed on at least 2 occasions for a period of at least 3 months, irrespective of the underlying cause and on the basis

    1. an estimated or measured glomerular filtration rate <60 mL/min/1.73 m2 and/or
    2. evidence of kidney damage (albuminuria, proteinuria, haematuria after exclusion of urological causes, or structural abnormalities on kidney imaging tests)

Exclusion Criteria:

* a subject who refuses to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
An occurrence of allopurinol-induced severe cutaneous adverse reaction | Before 3 months after initiation of allopurinol
  # Clinical presentations
  * Stevens-Johnson syndrome (SJS), SJS/Toxic epidermal necrolysis (TEN) overlap and TEN were diagnosed according to the range of detached surface area (< 10 %, 10-30 %, and > 30 %, respectively).
  * Drug rash with eosinophilia and systemic symptoms (DRESS) was diagnosed with the following criteria; Hospitalization, Reaction suspected to be drug-related Acute rash, Fever >38°C*, Enlarged lymph nodes at a minimum of 2 sites*, Involvement of at least 1 internal organ*, Blood count abnormalities*, Lymphocytes above or below normal limits, Eosinophils above the laboratory limits, Platelets below the laboratory limits [Three out of four asterisked (*) criteria are required for making the diagnosis.]

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea